CLINICAL TRIAL: NCT06898593
Title: Enhancing Engagement by Integrating Goals and Concerns That Matter to Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Dartmouth College (Other)
Responsible Party: Principal Investigator, Anna Tosteson, Principal Investigator, Trustees of Dartmouth College
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00033019 | STUDY02002511; 1UM1TR004772-01 (NIH)
Record Dates: First submitted 2025-03-14; First posted 2025-03-27 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-04

CONDITIONS: Anxiety Disorders; Depression Disorders
Keywords: Collaborative Care Model; pre-visit questionnaire; dashboard; clinical decision support system; Depression; Anxiety; integrated behavioral health and primary care
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Dashboard Systems

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster-randomized controlled trial (3 steps of 2 clinics each)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinical Decision Support System (Experimental): Collaborative care model, with a clinical decision support system (CDSS) which includes an enhanced pre-visit questionnaire and dashboard to visualize patient-reported information and clinical information.
  Interventions: Behavioral: Collaborative care model with clinical decision support system
- Collaborative care model (usual care) (Active Comparator): Standard collaborative care model of integrated behavioral health.
  Interventions: Behavioral: Collaborative care model

INTERVENTIONS:
Behavioral: Collaborative care model with clinical decision support system — A new patient-level clinical decision support system (CDSS) will include enhancing the existing pre-visit questionnaire to capture patient-reported goals and concerns, and displaying pre-visit questionnaire responses and clinical information within a patient-level dashboard in the electronic health record (EHR) for use by clinicians and patients.
  Other Names: dashboard; pre-visit questionnaire
  Arms: Clinical Decision Support System
Behavioral: Collaborative care model — Collaborative care model of integrated behavioral health and primary care.
  Arms: Collaborative care model (usual care)

SUMMARY:
The goal of this clinical trial is to learn if adding patients' goals and concerns to measurement-based collaborative care can tailor care and provide a more holistic view of treatment, thereby improving engagement in care among adult patients receiving collaborative care. The main questions it aims to answer are:

* Does using a clinical decision support system (which includes an enhanced pre-visit questionnaire and patient-level dashboard) improve patient engagement in the collaborative care model?
* Does using a clinical decision support system improve patient and clinician satisfaction with care?

Researchers will compare the enhanced collaborative care with traditional collaborative care.

Patient participants will complete pre-visit questionnaires before their collaborative care appointments. Responses will be viewed by the clinician and/or patient in a visual dashboard inside the electronic health record.

DETAILED DESCRIPTION:
Dartmouth Health (DH) has implemented the evidence-based Collaborative Care Model (CoCM) of integrated behavioral health in primary care.

CoCM includes (a) an initial behavioral health assessment with validated patient-reported outcomes, including the Patient Health Questionnaire (PHQ-9) and Generalized Anxiety Disorder (GAD-7) scale, (b) joint care planning and treatment with pharmacotherapy and/or psychotherapy, (c) monitoring using a registry to track treatment and patient-reported outcomes, and (d) caseload review with a psychiatric consultant.

There are several limitations associated with CoCM, including loss of patients between referral and treatment, failure to complete CoCM, and a limited ability to monitor for post-treatment relapse in depressive symptoms. These limitations are associated with low motivation to engage in BH services and patient perceptions that providers cannot accommodate their needs.

The scientific premise of the project is that structured collection and use of personalized treatment goals and concerns will improve patient engagement with CoCM, extending service impact. This study will highlight patient priorities for healthcare services to the CoCM team and will overcome clinical translational science challenges associated with patients' goals and concerns being neither fully documented nor available to support care, improvement, and research.

Enhancing patient-generated data collected through CoCM (e.g., PHQ-9; GAD-7) with patients' goals and concerns will reduce barriers to engagement in BH services by overcoming patient perceptions that services are misaligned with needs. Previous studies demonstrate that agenda setting processes that elicit priorities can improve clinicians' understanding of patients' concerns, increase patients' perceptions that what matters most is heard and incorporated into care plans, and increase likelihood of patients adhering to treatment recommendations.

Clinicians and patient stakeholders will use human-centered co-design principles to (a) enhance the existing CoCM pre-visit questionnaire (PVQ) to capture patient-reported goals and concerns, and (b) build a patient-level clinical decision support system (CDSS) that visualizes PVQ responses and clinical information within the electronic health record (EHR) for in-visit use by clinicians and patients. PVQs will support the patient in defining their visit agenda and providing an opportunity to align care with their immediate psychosocial and clinical needs. PVQs will be configured in Epic's MyChart® patient portal, allowing for completion at home prior to the visit or with a tablet upon clinic check-in. PVQ responses will be directly imported via a smart phrase into a clinical note template that clinicians can edit during the visit, reducing documentation burden and complexity. The care plan will be based on joint clinician and patient input and be available to the patient in the patient portal after the visit.

Intervention rollout will involve coaching CoCM care managers to use the CDSS following an established process. This will include a quality improvement curriculum to optimize use of the CDSS within clinical workflows and to incorporate patient preferences into decision-making. Training and support will be provided to care managers via monthly sessions informed by monitoring and feedback to assess and resolve challenges.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the Collaborative Care Model (CoCM) at Dartmouth Health

Exclusion Criteria:

* Patients not enrolled in the Collaborative Care Model (CoCM) at Dartmouth Health

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2448 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Engagement | From enrollment in CoCM to discharge from CoCM, approximately 3-4 months.
  The primary outcome measure targeted is increased Collaborative Care Model (CoCM) engagement as measured by the proportion of CoCM patients with 2 or more Patient Health Questionnaire (PHQ-9)/Generalized Anxiety Disorder (GAD-7) assessments completed.
Patient and clinician satisfaction and barriers/facilitators to implementation | From enrollment in CoCM to discharge from CoCM, approximately 3-4 months.
  Qualitative data collected through semi-structured interviews.

SECONDARY OUTCOMES:
Practice-level communication: Shared decision-making | Approximately 1 month following enrollment in CoCM
  Practice-level communication will be assessed using the collaboRATE measure of shared decision making. The collaboRATE survey includes three questions, rated from 0 (no effort was made) to 4 (every effort was made). Responses will be scored using the Top Score approach which excludes cases where a response to one or more of the collaboRATE questions is missing. Each encounter is coded as either '1', if the response to all three collaboRATE items was 4, or '0' if the response to any of the three collaboRATE items was less than 4. The percentage of all encounters that were coded as '1' is the collaboRATE Score. Higher scores represent more shared decision making.
Patient experience: Communication | Approximately 1 month following enrollment in CoCM
  Communication will be assessed using the "Communication with Mental Health Counselor" composite measure from the CAHPS Outpatient Mental Health Survey, which includes two questions: "In the last 6 months, how often did your main mental health counselor listen carefully to you? In the last 6 months, how often did your main mental health counselor show respect for what you had to say?" (Response options: never, sometimes, usually, always).
  The score for the composite measure is equal to the mean of the proportion of responses (excluding missing data) in each response category across the items in the composite, where the numerator is the number of people responding "always" and the denominator for each question is the total number of responses. Higher scores indicate higher quality communication.
Patient experience: Goal setting | Approximately 1 month following enrollment in CoCM
  Goal setting will be assessed using a single question from the CAHPS Outpatient Mental Health Survey: "In the last 6 months, how much did your main mental health counselor consider what is important to you when setting the goals for treatment?" (Response options: not at all, a little, some, a lot).
  The score is equal to the proportion of responses (excluding missing data) who indicate the top answer "a lot", divided by the total number of responses. Higher proportions indicate higher goal setting.
Treatment response: Depression | From enrollment in CoCM to discharge from CoCM, approximately 3-4 months.
  Change in depressive symptoms will be determined based on the scores obtained from the Patient Health Questionnaire-9 (PHQ-9). The total score can range from 0 to 27. Higher scores indicate greater severity of depression.
Treatment response: Anxiety | From enrollment in CoCM to discharge from CoCM, approximately 3-4 months.
  Change in anxiety symptoms will be determined based on scores obtained from the 7-item General Anxiety Disorder (GAD-7) scale. The total score can range from 0 to 21. Higher scores indicate greater severity of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Tosteson, ScD, Principal Investigator — Dartmouth College
Locations (6):
- United States (6):
  - Dartmouth Hitchcock Concord Family Medicine, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Dartmouth-Hitchcock Heater Road Internal Medicine, Lebanon, New Hampshire
  - Dartmouth Hitchcock Manchester Family Practice, Manchester, New Hampshire
  - Dartmouth Hitchcock Nashua Family Practice, Nashua, New Hampshire
  - Dartmouth Hitchcock Nashua General Internal Medicine, Nashua, New Hampshire

IPD SHARING:
Plan to Share IPD: No
IPD falls under patient protected health information (PHI).

REFERENCES:
- [Background] Barr PJ, Thompson R, Walsh T, Grande SW, Ozanne EM, Elwyn G. The psychometric properties of CollaboRATE: a fast and frugal patient-reported measure of the shared decision-making process. J Med Internet Res. 2014 Jan 3;16(1):e2. doi: 10.2196/jmir.3085. PMID 24389354
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Basch E, Barbera L, Kerrigan CL, Velikova G. Implementation of Patient-Reported Outcomes in Routine Medical Care. Am Soc Clin Oncol Educ Book. 2018 May 23;38:122-134. doi: 10.1200/EDBK_200383. PMID 30231381
- [Background] Oliver BJ, Nelson EC, Kerrigan CL. Turning Feed-forward and Feedback Processes on Patient-reported Data into Intelligent Action and Informed Decision-making: Case Studies and Principles. Med Care. 2019 May;57 Suppl 5 Suppl 1:S31-S37. doi: 10.1097/MLR.0000000000001088. PMID 30985594
- [Background] Tse CS, Van Citters AD, Ricci B, Freundlich NZ, Lee M, Shah SA, Melmed GY, Siegel CA, van Deen WK; IBD Qorus. Identifying and Predicting the Goals and Concerns Prioritised by Individuals with Inflammatory Bowel Disease. J Crohns Colitis. 2022 Mar 14;16(3):379-388. doi: 10.1093/ecco-jcc/jjab142. PMID 34350943
- [Background] Van Citters AD, Holthoff MM, Kennedy AM, Melmed GY, Oberai R, Siegel CA, Weaver A, Nelson EC. Point-of-care dashboards promote coproduction of healthcare services for patients with inflammatory bowel disease. Int J Qual Health Care. 2021 Nov 29;33(Supplement_2):ii40-ii47. doi: 10.1093/intqhc/mzab067. PMID 34849970
- [Background] Boudreau DM, Capoccia KL, Sullivan SD, Blough DK, Ellsworth AJ, Clark DL, Katon WJ, Walker EA, Stevens NG. Collaborative care model to improve outcomes in major depression. Ann Pharmacother. 2002 Apr;36(4):585-91. doi: 10.1345/aph.1A259. PMID 11918503
- See also: CAHPS Outpatient Mental Health Survey — https://www.ahrq.gov/cahps/surveys-guidance/mental-health/index.html
- See also: Patient Health Questionnaire-9 instrument — https://www.mdcalc.com/calc/1725/phq9-patient-health-questionnaire9
- See also: General Anxiety Disorder-7 instrument — https://www.mdcalc.com/calc/1727/gad7-general-anxiety-disorder7